CLINICAL TRIAL: NCT03214536
Title: Erector Spine Block in Patients Undergoing Back Surgery, Observational Feasibility Trial of the Effect on Postoperative Pain-scores and Opioid Consumption
Brief Title: Erector Spine Block for Back Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Dr M. B. Breebaart, principal investigator, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC nr 17/09/097
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Spine Disease; Regional Anaesthesia
Keywords: spine surgery; regional anaesthesia; opioid consumption; acute postoperative pain
MeSH Terms: conditions — Spinal Diseases; Pain, Postoperative | interventions — Ropivacaine; Anesthesia

STUDY DESIGN:
Intervention Model Description: observational feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- erector spinae block (Experimental): bilateral erector spine block with 20 ml 0,375% ropivacaine
  Interventions: Procedure: erector spinae block; Drug: Ropivacaine; Procedure: Spine surgery; Procedure: anesthesia

INTERVENTIONS:
Procedure: erector spinae block — bilateral injection of local anaesthetic between the erector spinae muscle and the transverse process
Drug: Ropivacaine — injection of 20 ml ropivacaine 0.375 % bilateral by erector spinae block
  Other Names: naropin
Procedure: Spine surgery — Surgery of lumbar spine
Procedure: anesthesia — general anesthesia

SUMMARY:
In spine surgery postoperative pain can often be severe and difficult to treat.With the use of ultrasound, the performance of plane blocks and other techniques like root blocks, facet infiltration have become possible without the use of either unreliable " pop-techniques" or the use of x-ray.The erector spinae block was recently described as a safe and simple and safe technique for neuropathic pain and acute post surgical pain, with effect on the dorsal rami of the spinal nerves and with promising results. In this observational pilot study we want to test the influence of these to blocks on the postoperative pain and opioid consumption after spine fusion.

DETAILED DESCRIPTION:
In 10-15 patients undergoing back surgery (laminectomy or back surgery with lumbar pedicle screw placement or revision back surgery), will be asked to give informed consent to receive a bilateral lumbar erector spinae block before surgery. In this population it will be clear after 10-15 patients if there is a beneficial effect since these patients normally require a substantial amount of postoperative opioids because of significant postoperative pain.

The blocks will be performed by experts in the field of ultrasound guided locoregional anaesthesia in a separate block room with ultrasound after placement of an iv line and application of standard monitoring (ECG, NIBP, saturation)

Description of block performance according to Chinn et al but at a lumbar level:

The patient will be placed in the lateral or sitting position. With a curve array probe or a high frequency linear probe, depending on the BMI of the patient, will be placed in a longitudinal position 2-3 cm lateral of the vertebral column. The transverse processes of the vertebrae at the (mid) level of surgery, the erector spinae muscle and the psoas muscle are identified. Depending on the depth a 5 or 8 cm 22 G ultrasound needle (pajunk) will be inserted in an in plane technique in a cephalad to caudad direction until bone contact with the top of the transverse process is reached. After slight retraction of the needle, 20 ml of ropivacaine 0,375% will be injected behind the erector spinae muscle. The same procedure will be repeated on the contralateral side.

Sensory loss of the posterior dermatomes and dermatomes of the anterior roots of the spinal nerves (lumbar plexus, upper leg) will be tested Motor function of the legs will be evaluated with a Bromage (0-3) score.

General anaesthesia will then be induced in a standardized way with propofol, sufentanyl and rocuronium. The maintenance of anaesthesia and the procedure will be performed according to protocol.

After surgery analgesia will be provided with nsaid when applicable and 1000 mg paracetamol IV 4 times daily combined with a PCA (patient controlled analgesia) pump depending on the site:

* AZ klina protocol: PCA piritramide/dhbp pump: 0ml/h, 2 mg bolus, 20 minutes lockout
* UZA protocol: Morphine/dhbp pump: 0ml/h 1 mg bolus, 8minutes lock out) and Pain scores (NRS, 0=no pain 10= worst pain ever), will be tested on the post anesthesia care unit every hour and according to hospital postoperative protocol at the ward during the fist 24 hours.

The amount and frequency of the opioid usage of the first 24 hours will be extracted out of the PCA pump. In patients without a block, opioid consumption is mostly expected between 25-40 mg morphine/24h (loading dose excluded) according to weight. We expect to see a substantial decrease (at least 50 %) in opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for laminectomy or back surgery with lumbar pedicle screw placement or revision back surgery

Exclusion Criteria:

* patient refusal, bleeding disorder, infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-25 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
24 hour opioid consumption | 24 hours from injection ( T0)
  cumulative opioid consumption first 24 hours after block performance

SECONDARY OUTCOMES:
sensory block | 30 minutes after block performance
  loss of cold sensation of anterior and posterior roots of lumbar spinal nerve dermatomes
motor block | 30 minutes after block performance
  motor function of legs by Bromage scale
pain scores | 24 postoperative at regular intervals
  numeric rating scores postoperative pain ( 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: margaretha breebaart, PhD, Principal Investigator — University Hospital, Antwerp
Locations (2):
- Belgium (2):
  - AZ KLina, Brasschaat, Antwerp
  - University Hospital Antwerp, Edegem, Antwerp

IPD SHARING:
Plan to Share IPD: Undecided